CLINICAL TRIAL: NCT00675337
Title: The Effect of Infant Placement at Delivery on Iron Stores in Early Infancy: A Pilot Study
Brief Title: Effect of Infant Placement on Iron Stores in Infancy: A Pilot Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Davison, James, D.O. (Individual)
Responsible Party: James M. Davison, DO, Warren General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: wghjmd1
Record Dates: First submitted 2008-05-07; First posted 2008-05-09 (Estimated); Last update posted 2008-12-31 (Estimated); Status verified 2008-12

CONDITIONS: Iron Deficiency; Anemia
Keywords: iron stores; anemia; iron deficiency; infancy; placental transfusion; iron deficiency in infancy; anemia in infancy; placement of neonate
MeSH Terms: conditions — Iron Deficiencies; Anemia; Fetofetal Transfusion

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- perineum (Active Comparator): infants maintained at the level of the perineum until umbilical cord clamping
  Interventions: Procedure: perineum maintained
- abdomen (Experimental): infants placed on the maternal abdomen prior to cord clamping
  Interventions: Procedure: abdominal placement

INTERVENTIONS:
Procedure: perineum maintained — infants maintained at the level of the perineum until umbilical cord clamping
  Arms: perineum
Procedure: abdominal placement — infants placed on the maternal abdomen prior to umbilical cord clamping
  Arms: abdomen

SUMMARY:
This is a pilot study designed to assess the safety of placing an infant on the mother's abdomen at the time of delivery, prior to clamping the umbilical cord and the effect of placing the infant on the mother's abdomen on the infant's iron stores. It is possible that placing the infant on the mother's abdomen (above the placenta) may lower the infant's iron stores during early infancy.

ELIGIBILITY:
Inclusion Criteria:

* healthy pregnant women
* 37 - 42 weeks of gestation
* vaginal delivery
* prenatal care initiated prior to 20 weeks of gestation

Exclusion Criteria:

* maternal diabetes
* intrauterine growth restriction
* hypertensive disorders of pregnancy
* chronic hypertension requiring medical therapy
* Apgar score less than 7 at 5 minutes
* unusual bleeding prior to delivery
* alloimmunization
* maternal hemoglobinopathy
* need for immediate infant resuscitation preventing adherence to protocol

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-06; Primary Completion 2008-12 (Actual); Study Completion 2009-04 (Estimated)

PRIMARY OUTCOMES:
serum ferritin level at 4 months of age | 4 months

SECONDARY OUTCOMES:
blood parameters (hemoglobin and hematocrit) | 2 months and 4 months
serum ferritin at 2 months | 2 months
blood parameters (hemoglobin and hematocrit) at 24 hrs of age | 24 hrs.

CONTACTS AND LOCATIONS:
Overall Officials: James M Davison, DO, Principal Investigator — Warren General Hospital; Sunny A Thomas, MD, Principal Investigator — Warren General Hospital

REFERENCES:
- [Background] Lozoff B, Beard J, Connor J, Barbara F, Georgieff M, Schallert T. Long-lasting neural and behavioral effects of iron deficiency in infancy. Nutr Rev. 2006 May;64(5 Pt 2):S34-43; discussion S72-91. doi: 10.1301/nr.2006.may.s34-s43. PMID 16770951
- [Background] Lozoff B, Georgieff MK. Iron deficiency and brain development. Semin Pediatr Neurol. 2006 Sep;13(3):158-65. doi: 10.1016/j.spen.2006.08.004. PMID 17101454
- [Background] Grant CC, Wall CR, Brewster D, Nicholson R, Whitehall J, Super L, Pitcher L. Policy statement on iron deficiency in pre-school-aged children. J Paediatr Child Health. 2007 Jul-Aug;43(7-8):513-21. doi: 10.1111/j.1440-1754.2007.01128.x. PMID 17635678
- [Background] Beard J. Recent evidence from human and animal studies regarding iron status and infant development. J Nutr. 2007 Feb;137(2):524S-530S. doi: 10.1093/jn/137.2.524S. PMID 17237340
- [Background] McCann JC, Ames BN. An overview of evidence for a causal relation between iron deficiency during development and deficits in cognitive or behavioral function. Am J Clin Nutr. 2007 Apr;85(4):931-45. doi: 10.1093/ajcn/85.4.931. PMID 17413089
- [Background] Burden MJ, Westerlund AJ, Armony-Sivan R, Nelson CA, Jacobson SW, Lozoff B, Angelilli ML, Jacobson JL. An event-related potential study of attention and recognition memory in infants with iron-deficiency anemia. Pediatrics. 2007 Aug;120(2):e336-45. doi: 10.1542/peds.2006-2525. PMID 17671043
- [Background] Walter T. Effect of iron-deficiency anemia on cognitive skills and neuromaturation in infancy and childhood. Food Nutr Bull. 2003 Dec;24(4 Suppl):S104-10. doi: 10.1177/15648265030244S207. PMID 17016952
- [Background] Levy T, Blickstein I. Timing of cord clamping revisited. J Perinat Med. 2006;34(4):293-7. doi: 10.1515/JPM.2006.056. PMID 16856818
- [Background] Ceriani Cernadas JM, Carroli G, Pellegrini L, Otano L, Ferreira M, Ricci C, Casas O, Giordano D, Lardizabal J. The effect of timing of cord clamping on neonatal venous hematocrit values and clinical outcome at term: a randomized, controlled trial. Pediatrics. 2006 Apr;117(4):e779-86. doi: 10.1542/peds.2005-1156. Epub 2006 Mar 27. PMID 16567393
- [Background] Hutton EK, Hassan ES. Late vs early clamping of the umbilical cord in full-term neonates: systematic review and meta-analysis of controlled trials. JAMA. 2007 Mar 21;297(11):1241-52. doi: 10.1001/jama.297.11.1241. PMID 17374818
- [Background] Yao AC, Lind J. Effect of gravity on placental transfusion. Lancet. 1969 Sep 6;2(7619):505-8. doi: 10.1016/s0140-6736(69)90213-x. No abstract available. PMID 4184835
- [Background] Grisaru D, Deutsch V, Pick M, Fait G, Lessing JB, Dollberg S, Eldor A. Placing the newborn on the maternal abdomen after delivery increases the volume and CD34 cell content in the umbilical cord blood collected: an old maneuver with new applications. Am J Obstet Gynecol. 1999 May;180(5):1240-3. doi: 10.1016/s0002-9378(99)70623-x. PMID 10329884
- [Background] Pafumi C, Zizza G, Russo A, Farina M, Pernicone G, Bandiera S, Giardina P, Mangiafico L, Mancari R, Maggi I, Calogero AE, Cianci A. Placing the newborn on the maternal abdomen increases the volume of umbilical cord blood collected. Clin Lab Haematol. 2001 Dec;23(6):397-9. doi: 10.1046/j.1365-2257.2001.00377.x. PMID 11843888
- [Background] Yao AC, Lind J. Placental transfusion. Am J Dis Child. 1974 Jan;127(1):128-41. doi: 10.1001/archpedi.1974.02110200130021. No abstract available. PMID 4588934
- [Background] Mercer JS, Nelson CC, Skovgaard RL. Umbilical cord clamping: beliefs and practices of American nurse-midwives. J Midwifery Womens Health. 2000 Jan-Feb;45(1):58-66. doi: 10.1016/s1526-9523(99)00004-5. PMID 10772736
- [Background] Siddappa AM, Rao R, Long JD, Widness JA, Georgieff MK. The assessment of newborn iron stores at birth: a review of the literature and standards for ferritin concentrations. Neonatology. 2007;92(2):73-82. doi: 10.1159/000100805. Epub 2007 Mar 14. PMID 17361090
- [Background] Beard JL, Murray-Kolb LE, Rosales FJ, Solomons NW, Angelilli ML. Interpretation of serum ferritin concentrations as indicators of total-body iron stores in survey populations: the role of biomarkers for the acute phase response. Am J Clin Nutr. 2006 Dec;84(6):1498-505. doi: 10.1093/ajcn/84.6.1498. PMID 17158435